CLINICAL TRIAL: NCT02293031
Title: Clinical Trial of Safety and Efficacy of the Medical Item Collagen Plates With Hydroxyapol Inducing Angiogenesis, "Nukleostim", for Bone Tissue Regeneration
Brief Title: Gene-activated Matrix for Bone Tissue Repair in Maxillofacial Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: NextGen Company Limited (Industry)
Collaborators: Burnasyan Federal Medical Biophysical Center (Other Government); Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU-NextGen-20-01-2013
Record Dates: First submitted 2014-11-11; First posted 2014-11-18 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2016-03

CONDITIONS: Maxillofacial Bone Defects; Alveolar Bone Atrophy; Jaw Fractures; Maxillofacial Bone Deformities; Bone Neoplasm, Benign; Disorders of Teeth and Jaw
Keywords: maxillofacial bone defects; alveolar ridge atrophy; gene-activated matrix; VEGF gene; DNA plasmid; bone gene therapy
MeSH Terms: conditions — Alveolar Bone Loss; Jaw Fractures; Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gene-activated matrix "Nucleostim" (Experimental): Implantation of gene-activated matrix "Nucleostim" into the bone defects or sites of bone atrophy
  Interventions: Device: Gene-activated matrix "Nucleostim"

INTERVENTIONS:
Device: Gene-activated matrix "Nucleostim" — Gene-activated matrix "Nucleostim" is bone graft substitute consisting of collagen-hydroxyapatite composite scaffold and DNA plasmids with gene encoding vascular endothelial grothw factor (VEGF-A165) in concentration 100-120 ng/mg which is an active substance of gene-therapeutic drug "Neovasculgen"®.

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of gene-activated matrix ("Nucleostim") for regeneration of bone tissue in maxillofacial area. Patients with congenital and acquired maxillofacial defects (sockets of extracted teeth, bone defects after injuries, surgeries, excision of benign neoplasms and pseudotumors, etc.) or alveolar bone atrophy will be included into the study.

DETAILED DESCRIPTION:
All patients enrolled into the study will receive standard surgery procedures indicated in accordance with medical care standards for the certain disease. Maxillofacial bone defects (formed after injuries, surgeries, excision of benign neoplasms and pseudotumors, teeth extraction, etc.) or areas of alveolar bone atrophy will be the filled by gene-activated matrix "Nucleostim". Safety and efficacy of implanted osteoplastic material will be assessed by physical examination, comprehensive laboratory tests, X-ray examination within 60 days after operation.

ELIGIBILITY:
Inclusion Criteria:

* obtained voluntary informed consent for participation in the clinical study;
* congenital and acquired maxillofacial bone defects (sockets of extracted teeth, bone defects after injuries, surgeries, excision of benign neoplasms and pseudotumors, etc.) or alveolar bone atrophy.

Exclusion Criteria:

* not able or unwilling to give voluntary informed consent for the study or follow requirements of the clinical study;
* decompensated chronic visceral diseases;
* clinically significant laboratory abnormalities;
* HIV, HBV and HCV antibodies in serum;
* alcohol consumption within 4 days prior the study;
* history of drug addiction;
* participation in other clinical studies (or administration of study products) within 3 months prior the study;
* conditions limiting study compliance (dementia, psycho-neurological diseases, drug addiction, alcoholism, etc.);
* malignancies including post-surgical period with chemo- and (or) radiation therapy);
* vascular malformations;
* pregnancy or lactation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Quantity of newly-formed bone tissue in the field of gene-activated matrix implantation | 60 days
  To determine the quantity of newly-formed bone tissue the morphometric parameters of regenerate will be measured on CT scan using special tools ("ROI", region of interest, etc.)
  The morphometric parameters of bone regenerate include:
  * average density (in HU);
  * size (length, width, height) and volume.

SECONDARY OUTCOMES:
Pain scores on the visual analog scale | 60 days
Surgical failure rate | 60 days
Adverse Events | 60 days
Edema scores on the 0-10 Numeric Rating Scale | 60
  Level of edema at the surgical site will be assessed by physician using 0-10 Numeric Rating Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Yu Drobyshev, MD, PhD, DSc, Principal Investigator — Moscow State University of Medicine and Dentistry
Locations (2):
- Russia (2):
  - Burnasyan Federal Medical Biophysical Center, Moscow
  - Moscow State University of Medicine and Dentistry, Moscow

REFERENCES:
- [Background] Bozo I.Y., Deev R.V., Drobyshev A.Y., D. Galetskiy D.V., Isaev A.A. Gene technologies in maxillofacial surgery: development of gene-activated bone grafts. International Journal of Oral and Maxillofacial Surgery 42(10): 1179-1180, 2013
- [Background] Deev R.V., Drobyshev A.Y., Bozo I.Y., Isaev A.A. Angiogenic non-viral gene transfer: from ischemia treatment to bone defects repair. J Tissue Eng. Regen. Med. 8 (Suppl. 1): 64-65, 2014
- [Background] Deev RV, Bozo IIa, Mzhavanadze ND, Nersesian EG, Chukhralia OV, Shval'b PG, Cherviakov IuV, Staroverov IN, Kalinin RE, Voronov DA, Gavrilenko AV, Isaev AA. [Efficacy of using VEGF165 gene in comprehensive treatment of patients with stage 2A-3 lower limb chronic ischaemia]. Angiol Sosud Khir. 2014;20(2):38-48. Russian. PMID 24961325
- [Result] Bozo IY, Deev RV, Drobyshev AY, Isaev AA, Eremin II. World's First Clinical Case of Gene-Activated Bone Substitute Application. Case Rep Dent. 2016;2016:8648949. doi: 10.1155/2016/8648949. Epub 2016 Nov 7. PMID 27891264